CLINICAL TRIAL: NCT06971835
Title: Assessment of Safety and Clinical Effectiveness of Induce NMP® in Degenerative Spine Surgery: A Prospective 2-Year Registry
Brief Title: INDUCE: A Prospective 2-Year Spine Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Red Rock Regeneration Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-NMP-009
Record Dates: First submitted 2025-04-23; First posted 2025-05-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Subjects Treated With NMP as Part of Their Spine Surgery; Degenerative Disc Disease (DDD)
Keywords: degenerative spine; NMP; Induce
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects treated on-label with NMP as part of their spine surgery.: Subjects implanted on-label with NMP in at least one vertebral level in the cervical (C1-C7) or lumbar (L1-S1) spine as part of their surgery.
  Interventions: Device: NMP

INTERVENTIONS:
Device: NMP — The study product is Induce Biologics NMP Fibers and NMP Micro Particulates however, this is observational research that involves standard of care.
  NMP is regulated as a human cellular or tissue-based product (HCT/P) under section 361 of the Public Health Service (PHS) Act and in 21 CFR Part 1271. Under this regulation it did not require clinical evaluation before it could be used commercially. It is indicated for use "as a bone void filler for filling voids and gaps in the skeletal system that are not intrinsic to the stability of the boney structure.

SUMMARY:
The primary objective of this prospective, observational registry study is to evaluate the safety and effectiveness of Natural Matrix Protein® (NMP®) when used to promote fusion in the cervical or lumbar spine.

The secondary objective is to assess patient reported outcomes following the use of NMP in the treatment of the spine.

DETAILED DESCRIPTION:
This is a multicenter, observational, prospective registry study of up to 1,000 patients across a maximum of 10 US sites. All subjects who meet study entrance criteria and planned to be treated with NMP Fibers and/or Micro Particulates as part of their cervical or lumbar spinal surgery will be invited to participate in the study.

PRIMARY ENDPOINTS

* Safety - freedom from product-related serious adverse events and subsequent surgical interventions at the treated level(s)
* Effectiveness - presence of fusion as measured by x-rays and if available CT.

SECONDARY ENDPOINTS

Beyond the primary endpoints, the following data may be collected and analyzed including, but not limited to, the following variables:

* Baseline demographics and medical history
* Duration of hospitalization
* Operative time
* Estimated blood loss
* Neurological status
* Subject patient reported outcomes as applicable including, but not limited to:

  * Oswestry Disability Index (ODI)/ Neck Disability Index (NDI)
  * Visual Analog Scale (VAS) Pain
  * Veteran Rand 12-Item Health Survey (VR-12)

ELIGIBILITY:
Inclusion Criteria:

1. Implanted on-label with NMP in at least one vertebral level in the cervical (C1-C7) or lumbar (L1-S1) spine as part of their surgery
2. Total volume of bone graft or bone graft substitute used in index surgery must contain at least 50% NMP by volume per treated level, where NMP is mixed with other graft material.
3. Skeletally mature (age≥18 years of age)
4. Be willing to sign the study-specific informed consent document prior to index surgery

Exclusion Criteria:

1. Not willing to sign the study-specific informed consent document prior to index surgery
2. Use of allogenic growth factor extacts (i.e. OsteoFactor/ProteiOS) or cell based allografts as part of the index surgery (use of autograft or bone marrow aspirate (BMA) is allowed)
3. Use of rhBMP-2 (i.e. INFUSE) or synthetic peptide enhanced graft (i.e. iFactor) as part of the index surgery
4. Diagnosis of spinal deformity (greater than 20 degrees) or vertebral fracture including treated level
5. Unable to comply with postoperative standard of care imaging (e.g. pregnant or nursing female)
6. Did not complete baseline patient reported outcomes prior to index surgery
7. Incarcerated at the time of surgery or preoperative evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include a maximum of 10 US sites, covering a large geographic region, representing a diverse demographic cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Fusion | 6 month and 12 month post surgery, and 24 month post surgery
  Incidence of fusion at treated levels as measured by x-rays and if available CT, will be reported.
Serious Adverse Events and Subsequent Surgical Interventions | Through study completion, an average of 2 years.
  Incidence of serious adverse events (SAE) and subsequent surgical intervention (SSI) will be reported.

SECONDARY OUTCOMES:
Change in Pain | Baseline, 3 month, 6 months, 12 months, and 24 months postop
  Pain scores will be reported as assessed by Visual Analog Scale scores, (0-100mm) or Numeric Rating Scale (0-10) depending on institutions standard of care. Higher score indicates increased pain.
Change in Disability | Baseline, 3 month, 6 months, 12 months, and 24 months postop
  Disability improvement as measured by Oswestry Disability Index (ODI) or Neck Disability Index (NDI), as applicable, 0-100%. High score indicates increase disability.
Change in Quality of Life | Baseline, 3 month, 6 months, 12 months, and 24 months postop
  Improvement in qualify of life as measured by Veterans Rand-12, 0-100. High score indicates increase quality of life.

IPD SHARING:
Plan to Share IPD: No